CLINICAL TRIAL: NCT01125943
Title: Bevacizumab and Endothelium Dependent Vasodilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, G. Rongen, Prof dr. G. Rongen, Radboud University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BVZAch
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Hypertension; Cancer; Endothelial Dysfunction
MeSH Terms: conditions — Hypertension; Neoplasms | interventions — Acetylcholine; Nitroprusside; Bevacizumab

ARMS (2):
- Acetylcholine (Experimental): Intra-arterial infusion of acetylcholine in two increasing dosages during 5 minutes each during the intra-arterial infusion of bevacizumab
  Interventions: Drug: Acetylcholine; Drug: Bevacizumab
- Nitroprusside (Experimental): Infusion of two increasing dosages of nitroprusside during 5 minutes each during the continuous infusion of bevacizumab
  Interventions: Drug: Nitroprusside; Drug: Bevacizumab

INTERVENTIONS:
Drug: Acetylcholine — Intra-arterial infusion
  Arms: Acetylcholine
Drug: Nitroprusside — Intra arterial infusion
  Arms: Nitroprusside
Drug: Bevacizumab — Intra arterial infusion

SUMMARY:
The introduction of angiogenesis inhibitors has remarkably improved treatment of patients with several types of cancer. One of the most reported side effects of angiogenesis inhibitors is hypertension. In patients treated with bevacizumab, a monoclonal antibody against vascular endothelial growth factor, hypertension had an overall incidence up to 32%. The increase in blood pressure occurs early in treatment. The etiology of hypertension caused by treatment with angiogenesis inhibitors is unclear. Understanding the pathogenesis of this side effect is essential for optimal treatment with this class of drugs.

The primary objective is to explore the effect of bevacizumab infusion on endothelium-dependent vasodilation of forearm resistance arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 years old
2. Male
3. Results of serum glucose, lipids and creatinine should be within the laboratory's reference ranges.
4. Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.

Exclusion Criteria:

1. Documented history of sensitivity/idiosyncrasy to medicinal products or excipients.
2. History of or current abuse of drugs, alcohol or solvents.
3. History of malignant disease.
4. First degree relatives with a history of cancer before the age of 50
5. First degree relatives with a history of premature cardiovascular disease before the age of 50
6. Current use of medication.
7. Clinical evidence of cardiac or pulmonary disease
8. Hypertension ( systole >140mmHG, diastole >90mmHg)
9. Diabetes mellitus
10. Smoking
11. Any clinically relevant abnormality on ECG.
12. A history of thrombosis or first degree family members with a history of recurrent thrombosis
13. Inability to understand the nature and extent of the trial and the procedures required.
14. Previous participation in a study with bevacizumab

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Vasomotor response assessed by venous occlusion strain gauge plethysmography | 15 minutes
  Response to infusion of bevacizumab and/or acetylcholin or nitroprusside

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands